CLINICAL TRIAL: NCT07397351
Title: OPEN-LABEL, RANDOMIZED, MULTICENTER CLINICAL TRIAL TO EVALUATE THE CARDIOPROTECTIVE EFFECT, TO DETERMINE OPTIMAL DOSAGES AND DURATION OF INHALATION, AND TO CONFIRM THE CLINICAL SAFETY OF THE MEDICINAL PRODUCT AROXXEN® IN PATIENTS WHO HAVE UNDERGONE ELECTIVE PERCUTANEOUS CORONARY INTERVENTION WITH STENT IMPLANTATION (PHASE II)
Brief Title: OPEN-LABEL, RANDOMIZED, MULTICENTER PHASE II STUDY OF AROXXEN® INHALATION FOR CARDIOPROTECTION AFTER ELECTIVE PCI WITH STENT IMPLANTATION
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Research Institute of Geroprotective Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTARE25/II
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease; Myocardial Injury Associated With Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Patients receive inhalation of the investigational medicinal product Aroxxen® (composition variant 1) during and after elective percutaneous coronary intervention with stent implantation, according to the study protocol.
  Interventions: Drug: Aroxxen
- Group B (Experimental): Patients receive inhalation of the investigational medicinal product Aroxxen® (composition variant 2) during and after elective percutaneous coronary intervention with stent implantation, according to the study protocol.
  Interventions: Drug: Aroxxen
- Group C (No Intervention): Patients undergo elective percutaneous coronary intervention with stent implantation without additional inhalation of the investigational medicinal product.

INTERVENTIONS:
Drug: Aroxxen — Aroxxen® is an investigational medicinal product administered by inhalation during and after elective percutaneous coronary intervention in accordance with the study protocol.
  Arms: Group A; Group B

SUMMARY:
This is an open-label, randomized, multicenter Phase II clinical study designed to evaluate the cardioprotective effect, to determine the optimal dosages and duration of inhalation, and to assess the clinical safety of the medicinal product Aroxxen® in patients undergoing elective percutaneous coronary intervention (PCI) with stent implantation.

Patients who undergo elective PCI are at risk of myocardial injury associated with the procedure. The study aims to assess whether inhalation of Aroxxen®, administered during the procedure and after it, can reduce markers of myocardial damage and improve clinical outcomes, while maintaining an acceptable safety profile.

Eligible patients will be randomized to receive inhalation of Aroxxen® according to the study protocol or standard therapy without inhalation, depending on the assigned group. The study includes multiple centers and compares different dosing regimens and durations of inhalation in order to identify optimal treatment parameters.

Safety will be evaluated by monitoring adverse events, vital signs, and clinical laboratory parameters throughout the study period. The results of this study are intended to provide data on the safety and potential cardioprotective effects of Aroxxen® and to support further clinical development.

ELIGIBILITY:
1. Presence of coronary artery disease with stenosis of one or more coronary arteries requiring elective percutaneous coronary intervention for stent implantation (including patients with stable angina pectoris, Canadian Cardiovascular Society functional class II-IV, and patients with post-infarction or atherosclerotic cardiosclerosis with or without angina).
2. Clinically and/or hemodynamically significant coronary artery stenosis confirmed by coronary angiography, with an indication for percutaneous coronary intervention with stent implantation.
3. Age 50 to 80 years inclusive at the time of signing informed consent.
4. Baseline high-sensitivity troponin I within the laboratory reference range, excluding acute coronary syndrome.
5. Written voluntary informed consent obtained after the participant has received full information about the study objectives, methods, risks, and potential benefits.
6. Willingness and ability to comply with all study procedures and visits specified in the protocol.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incremental area under the concentration-time curve (iAUC) of high-sensitivity troponin I (hs-cTnI) | From baseline before the start of inhalation to 24 hours after the start of inhalation (with assessments at 4, 12, and 24 hours).
  The individual incremental area under the concentration-time curve (iAUC) of high-sensitivity troponin I is calculated for each participant based on serial venous blood measurements obtained at baseline before the start of inhalation and at 4 hours, 12 hours, and 24 hours after the start of inhalation.